CLINICAL TRIAL: NCT02515435
Title: Single Arm Phase II Clinical Trial to Investigate the Efficacy and Safety of Apatinib as a Single Agent in Advanced NSCLC Who Failed to at Least Two Lines Systemic Treatment, or Were Not Amendable to Receive the Second-line Standard Therapy
Brief Title: The Efficacy and Safety of Apatinib in Heavily Pretreated Advanced Non-squamous Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tongji University (Other)
Responsible Party: Principal Investigator, Caicun Zhou, Pro, Dr, Tongji University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FK1405
Record Dates: First submitted 2015-07-30; First posted 2015-08-04 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: apatinib; NSCLC; safety; efficacy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- apatinib single agent (Experimental): apatinib, single agent, 500mg or 750mg Qd po, continue until disease progression
  Interventions: Drug: apatinib single agent

INTERVENTIONS:
Drug: apatinib single agent — For those heavily treated non-squamous non-small cell lung cancer, treat with apatinib single agent, 500mg or 750mg Qd, p.o based on the status of patient, continue until disease progression, dose reduction was admitted
  Other Names: YN968D1

SUMMARY:
The development of anti-angiogenesis drugs has led to renewed enthusiasm in lung cancer treatments. Apatinib, also known as YN968D1, is a tyrosine kinase inhibitor which selectively inhibits the vascular endothelial growth factor receptor-2 (VEGFR-2) and also represents mild inhibition to PDGFR, c-Kit and c-src tyrosine kinases. It is an orally bioavailable, small molecule agent which is thought to inhibit VEGF-mediated endothelial cell migration and proliferation thus blocking blood vessel formation in tumor tissues. Previous studies have identified that apatinib was well tolerated at doses below 750mg daily. In phase I/II study, investigators reported an objective response rate of 68%. In a phase III trial conducted in advanced pretreated gastric cancer, the median overall survival was significantly prolonged in the apatinib group compared with placebo group. Thus, in this trial, the investigators aim to investigate the efficacy and safety of apatinib in previously treated advanced non-squamous non-small cell lung cancer.

DETAILED DESCRIPTION:
Observing the efficacy and safety of apatinib in heavily treated non-squamous non-small cell lung cancer.

Primary Outcome Measure: Objective Response Rate Secondary Outcome Measures: Progression free survival, overall survival, Side effects, Quality Of Life

ELIGIBILITY:
Inclusion Criteria:

1. Obtain of informed consent.
2. Aged 18 years and over.
3. Histologically or cytologically confirmed non-squamous non-small cell lung cancer.
4. World Health Organization (WHO) performance status (PS) of 0 to 2.
5. Measurable lesions as defined by RECIST criteria.
6. Life expectancy ≥12 weeks.
7. Progressed after at least two lines systemic treatment, or were not amendable to receive the current standard therapy

7. Organ functions normal, as defined below, within two weeks of randomization: Hb≥90g/L Absolute neutrophils count(ANC)≥1.5×109/L Platelets≥80×109/L Serum bilirubin≤2×ULN; Aspartate transaminase(AST) and alanine transaminase (ALT)≤2.5×ULN(≤5×ULN if liver metastases) Creatinine clearance≥45ml/min or Cr≤1.25×ULN 8. Females of child-bearing potential must have negative serum pregnancy test. Sexually active males and females (of childbearing potential) willing to practice contraception during the study.

Exclusion Criteria:

1. Squamous carcinoma (including adeno-squamous carcinoma), small cell lung cancer.
2. Newly diagnosed Central Nervous System (CNS) metastases that have not yet been definitively treated with surgery and/or radiation.
3. Tumor invade big vessels or close to big vessels (less than 5mm)
4. Obvious cavity or necrosis formed in the tumor
5. Uncontrolled hypertension
6. Myocardial ischemia or infarction more than stage II, cardiac insufficiency.
7. Abnormal coagulation (INR>1.5 or PT>ULN+4, or APTT>1.5 ULN), bleeding tendency or receiving coagulation therapy
8. Hemoptysis, more than 2.5ml daily
9. Thrombosis in 12 months, including pulmonary thrombosis, stoke, or deep venous thrombosis.
10. Unhealed bone fracture or wound for long time
11. Received big surgery, had bone fracture or ulcer in 4 weeks.
12. Urine protein≥++, or urine protein in 24 hours≥1.0g
13. Pregnant or lactating woman.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-01-01; Primary Completion 2016-08-01 (Actual); Study Completion 2017-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | tumor assessment every 2 cycles after the initiation of apatinib，up to 24 months
  To evaluate Objective response rate every 6-8 weeks after the initiation of apatinib.

SECONDARY OUTCOMES:
Progression free survival | 12 months
  PFS is evaluated in 24 months since the treatment began

OTHER OUTCOMES:
Overall survival | 12 months
  evaluated in the 24th month since the treatment began
side effects | 12 months
  evaluated in the 24th month since the treatment began according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Quality of life | 12 months
  evaluated in the 24th month since the treatment began

CONTACTS AND LOCATIONS:
Overall Officials: caicun zhou, MD,PhD, Principal Investigator — Shanghai Pulmonary Hospital, Tongji University
Locations (1):
- Department of Oncology, Shanghai pulmonary hospital, Shanghai, China

REFERENCES:
- [Derived] Wu F, Zhang S, Xiong A, Gao G, Li W, Cai W, Su C, Chen X, Zhou F, Zhao J, Ren S, Zhou C. A Phase II Clinical Trial of Apatinib in Pretreated Advanced Non-squamous Non-small-cell Lung Cancer. Clin Lung Cancer. 2018 Nov;19(6):e831-e842. doi: 10.1016/j.cllc.2018.06.002. Epub 2018 Jun 27. PMID 30026059